CLINICAL TRIAL: NCT01653626
Title: A Matched Pair Cluster-randomized Implementation Study to Measure the Effectiveness of an Intervention Package Aiming to Decrease Perinatal Mortality and Increase Institution-based Obstetric Care Among Indigenous Populations in Guatemala
Brief Title: A Study to Measure the Effectiveness of an Intervention Package Aiming to Decrease Perinatal Mortality and Increase Institution-based Obstetric Care Among Indigenous Populations in Guatemala
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Juan de Dios Guatemala (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Edgar Kestler, Director, World Health Organization
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: GUACTEK01
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: ¨Maternal Morbidity¨; ¨Perinatal Mortality¨
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- package (Experimental)
  Interventions: Other: package of 3 interventions

INTERVENTIONS:
Other: package of 3 interventions — Emergency Obstetric Care training, social marketing approach and link TBS with public sector services

SUMMARY:
A matched pair cluster-randomized trial of this intervention package will be conducted in four rural and indigenous districts (Huehuetenango, Quiche, Alta Verapaz and San Marcos) of the Republic of Guatemala, using the health clinic as the unit of randomization. No external intervention is planned for control facilities, although enhanced monitoring, surveillance and data collection will occur throughout the study in all facilities in the four districts.

The package includes 3 interventions: 1) To train health care professionals in emergency obstetric and perinatal care using an innovative high-fidelity, low-tech, in situ, multidisciplinary simulation training curriculum (PRONTO); 2) To design and implement a social marketing strategy that promotes institution-based delivery; and 3) To integrate the role of obstetric nurse and professional midwife in intervention communities to act as liaisons between traditional birth attendants (TBA) and public health units. A fourth, cross-cutting component involves ongoing analysis, monitoring, surveillance and evaluation to strengthen information systems and monitor perinatal outcomes throughout the two years of the study.

DETAILED DESCRIPTION:
Overall goal

To evaluate the impact of a package of three interventions aiming to increase institution-based delivery and improve emergency obstetric and neonatal care on perinatal mortality, in the four districts with the highest maternal mortality ratios in Guatemala.

Specific objectives

* Measure the impact of this intervention package on perinatal mortality rates.
* Measure the impact of this intervention package on the proportion of institution-based delivery among study facilities.
* Evaluate the processes and success of implementing this combined package of interventions by analyzing process indicators related to the intervention element designed to improve emergency obstetric and neonatal care (PRONTO: emergency obstetric and perinatal training program).

Primary outcome of interest:

1. Increase in the proportion of institutional deliveries in intervention vs. control clusters.
2. Decrease perinatal death rate in intervention vrs control clinics

ELIGIBILITY:
Inclusion Criteria:

* rural women
* indigenous
* poor
* Facilities at rural area
* Clinic attending vaginal deliveries

Exclusion Criteria:

* Facilities considered too close geographically to risk contamination of intervention to control facilities
* Clinics visits by pregnant women who present to intervention or control clinics for reasons other that an obstetric event
* Clinic or hospital visits by women who present to intervention or control clinics in the post partum period

Ages: 10 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
increase the proportion of institutional deliveries in intervention vs. control clusters | Up to 15 months

SECONDARY OUTCOMES:
Decrease perinatal death rate in intervention vs. control clinics | Up to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Edgar E Kestler, MD, Principal Investigator — CIESAR; Edgar E. Kestler, MD, Principal Investigator — CIESAR
Locations (1):
- Health Centers for vaginal deliveries (CAP), Departamento de San Marcos, Departamento de Guatemala, Guatemala

REFERENCES:
- [Derived] Walker DM, Holme F, Zelek ST, Olvera-Garcia M, Montoya-Rodriguez A, Fritz J, Fahey J, Lamadrid-Figueroa H, Cohen S, Kestler E. A process evaluation of PRONTO simulation training for obstetric and neonatal emergency response teams in Guatemala. BMC Med Educ. 2015 Jul 24;15:117. doi: 10.1186/s12909-015-0401-7. PMID 26206373
- [Derived] Kestler E, Walker D, Bonvecchio A, de Tejada SS, Donner A. A matched pair cluster randomized implementation trail to measure the effectiveness of an intervention package aiming to decrease perinatal mortality and increase institution-based obstetric care among indigenous women in Guatemala: study protocol. BMC Pregnancy Childbirth. 2013 Mar 21;13:73. doi: 10.1186/1471-2393-13-73. PMID 23517050